CLINICAL TRIAL: NCT02874118
Title: Search for Fragility Indicators Among People Aged 50+ With Chronic HIV Infection
Acronym: Visage 3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2011-41; 2011-A01679-32 (Other: Ansm)
Record Dates: First submitted 2016-08-17; First posted 2016-08-22 (Estimated); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Frail in HIV Population

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HIV Patient population over 50 years old (Experimental)
  Interventions: Behavioral: Fried scale for frailty assessement

INTERVENTIONS:
Behavioral: Fried scale for frailty assessement

SUMMARY:
The frailty and frail elderly was defined in 2001 by Fried as a physiological state of heightened vulnerability to external shocks. 5 criteria for classifying the elderly in 3 categories: frail, pre-frail and not frail. The prevalence of frailty in the general population was estimated to be 7%, 10% and 20% for over 65 years and 45% for over 85 years. This concept is explored in some chronic diseases, in order to prevent the loss of autonomy and tailor the treatment. In the carrier population of HIV, a North American retrospective study showed the frailty syndrome manifested as early as 10 years before, than in the general population. Furthermore various studies show in this specific population, increased incidence of diseases linked to age, suggesting an accelerated and premature aging.

objectives: The objective of this study is to determine the prevalence of frailty defined Fried syndrome in a population of subjects aged 50 and over Holders of chronic HIV infection.

ELIGIBILITY:
Inclusion Criteria:

* Patient with HIV and followed in the southeastern France area

Exclusion Criteria:

* In patient HIV infected patient
* HIV patient disabled (spastic)
* HIV infected for less than a year

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 510 (Actual)
Dates: Start 2012-09-26 (Actual); Primary Completion 2014-06-10 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
Number of frailed patient among the HIV population folloxed in southeastern France area | one year

CONTACTS AND LOCATIONS:
Overall Officials: Ureielle DESALBRES, Study Director — Assistance Publique Hôpitaux de Marseille; Nathalie PETIT, MD, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No